CLINICAL TRIAL: NCT05986318
Title: Reducing Respiratory Symptoms of Pulmonary Irradiation in Interstitial Lung Disease: A 2x2 Factorial Randomized Phase II Trial Testing N-Acetyl Cysteine and Dexamethasone
Brief Title: Reducing Respiratory Symptoms of Pulmonary Irradiation in Interstitial Lung Disease
Acronym: RESPIRE-ILD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Palma (Other)
Collaborators: London Health Sciences Centre (Other); Centre Hospitalier de l'Universite de Montreal (CHUM) (Unknown)
Responsible Party: Sponsor-Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RESPIRE-ILD
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer; Interstitial Lung Disease
Keywords: Pulmonary Irradiation; Radiation Therapy; N-Acetyl Cysteine; Dexamethasone; Radiation Pneumonitis
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases, Interstitial; Radiation Pneumonitis | interventions — Acetylcysteine; Dexamethasone; Adrenal Cortex Hormones; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NAC + Corticosteroids (Active Comparator): Participants will take 600 mg of active NAC orally, three times daily, for 60 days.
  Participants will also take 4 mg of active dexamethasone, orally, once daily for 10 days, then 2 mg, orally, once daily for 5 days, then 1 mg, orally, once daily for 5 days.
  All participants will be treated with radical pulmonary radiation therapy.
  Interventions: Dietary Supplement: N-Acetyl cysteine; Drug: Dexamethasone Oral; Radiation: Radiation Therapy
- Corticosteroids + NAC Placebo (Active Comparator): Participants will take 4 mg of active dexamethasone, orally, once daily for 10 days, then 2 mg, orally, once daily for 5 days, then 1 mg, orally, once daily for 5 days.
  Participants will also take matching NAC placebo orally, three times daily, for 60 days.
  All participants will be treated with radical pulmonary radiation therapy.
  Interventions: Drug: Dexamethasone Oral; Dietary Supplement: N-Acetyl cysteine Placebo; Radiation: Radiation Therapy
- NAC + Dexamethasone Placebo (Active Comparator): Participants will take 600 mg of active NAC orally, three times daily, for 60 days.
  Participants will also take matching dexamethasone placebo (4 mg for 10 days, then 2 mg for 5 days, then 1 mg for 5 days), orally, once daily.
  All participants will be treated with radical pulmonary radiation therapy.
  Interventions: Dietary Supplement: N-Acetyl cysteine; Drug: Dexamethasone Placebo; Radiation: Radiation Therapy
- NAC Placebo + Dexamethasone Placebo (Placebo Comparator): Participants will take matching NAC placebo orally, three times daily, for 60 days.
  Participants will also take matching dexamethasone placebo (4 mg for 10 days, then 2 mg for 5 days, then 1 mg for 5 days), orally, once daily.
  All participants will be treated with radical pulmonary radiation therapy.
  Interventions: Dietary Supplement: N-Acetyl cysteine Placebo; Drug: Dexamethasone Placebo; Radiation: Radiation Therapy

INTERVENTIONS:
Dietary Supplement: N-Acetyl cysteine — NAC capsules
  Other Names: NAC
  Arms: NAC + Corticosteroids; NAC + Dexamethasone Placebo
Drug: Dexamethasone Oral — Dexamethasone tablets
  Other Names: Corticosteroid
  Arms: Corticosteroids + NAC Placebo; NAC + Corticosteroids
Dietary Supplement: N-Acetyl cysteine Placebo — Matching placebo for NAC capsules
  Other Names: NAC Placebo
  Arms: Corticosteroids + NAC Placebo; NAC Placebo + Dexamethasone Placebo
Drug: Dexamethasone Placebo — Matching placebo for dexamethasone tablets
  Other Names: Corticosteroid Placebo
  Arms: NAC + Dexamethasone Placebo; NAC Placebo + Dexamethasone Placebo
Radiation: Radiation Therapy — All participants will receive radical pulmonary radiation therapy. Conventional techniques or stereotactic ablative radiotherapy will be used.

SUMMARY:
In this double-blind phase II randomized controlled trial, patients with lung cancer or ≤2 oligometastatic pulmonary lesions and a concomitant diagnosis of ILD who are planned for radical Radiation Therapy (RT) will be randomized using a 2 x 2 factorial design to oral N-acetylcysteine (NAC) versus placebo, and also to short course corticosteroids versus placebo.

DETAILED DESCRIPTION:
Radiation pneumonitis (RP) is the most common and main dose-limiting toxicity after thoracic RT. RP is characterized histologically by diffuse alveolar damage and acute vascular permeability induced by direct cytotoxic effect and oxidative stress, leading to the production of proinflammatory, profibrogenic and proangiogenic cytokines.

Patients with Interstitial Lung Disease (ILD) are at increased risk of developing lung cancer compared to the general population. Management of patients with lung cancer in the setting of a concomitant ILD is complex, as these patients are usually not good candidates for surgery or immunotherapy. In addition, patients with ILD, particularly fibrotic ILD, are also reportedly at increased risk of treatment-related toxicity from RT.

In the present study, investigators will test the following hypotheses:

1. The use of NAC with RT in patients with underlying ILD will lead to a clinically meaningful reduction in grade 2-5 dyspnea (as per Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).
2. The use of corticosteroids with RT in patients with underlying ILD will lead to a clinically meaningful reduction in grade 2-5 dyspnea (as per CTCAE version 5.0).

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer or 1-2 oligometastatic pulmonary lesions planned for radical intent radiotherapy [minimal Biologically Effective Does (BED) of 48 Gy10 (Gray) or biological equivalent].
* Pathologically (histologically or cytologically) proven diagnosis of cancer is not required, but strongly recommended.

  * If the risk of biopsy is unacceptable, pathologic confirmation is not required providing there is growth over time on Computed Tomography (CT) imaging and/or Fluorodeoxyglucose (FDG) avidity that is strongly suggestive of malignancy.
* Fibrotic Interstitial Lung Disease (ILD) of any subtype, as diagnosed by a respirologist and confirmed by central review
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Age ≥ 18
* Life expectancy > 6 months
* Patients are allowed to receive anti-fibrotic agents used in the treatment of Idiopathic Pulmonary Fibrosis (IPF) or non-IPF fibrotic ILD (e.g. nintedanib, pirfenidone) and/or corticosteroids, if those are part of their current ILD treatment regimen. Other immunosuppressive drugs such as mycophenolate, azathioprine, cyclophosphamide, and rituximab must be stopped for 2 weeks prior and 2 weeks after Radiation Therapy (RT).
* Concurrent standard chemotherapy is allowed where indicated. All other systemic therapies, including biologic targeted agents or immunotherapy, or any drugs with known radiosensitive effects, must be stopped for 2 weeks prior and 2 weeks after treatment.

Exclusion Criteria:

* Prior lung radiotherapy
* Current use of oral or intravenous corticosteroids
* Plans for the patient to receive other local therapy to the target lesion(s) while on this study, except at disease progression
* Any medical condition that could, in the opinion of the investigator, preclude radiotherapy or prevent follow-up after radiotherapy
* Pregnancy

  * If not pregnant, use of effective contraception methods for women of childbearing age is required which can include:

    * hormonal methods (e.g. oral, injected, implanted),
    * placement of an intrauterine device,
    * barrier methods (i.e. condoms),
    * sterilization of the partner (e.g. previous vasectomy)
    * abstinence
  * Women who become pregnant should stop taking NAC and/or dexamethasone and inform their study doctor.
  * Male participants should use adequate forms of birth control with their partners.
* Currently breastfeeding
* Current or recent use of NAC
* Contraindications to dexamethasone or N-Acetyl Cysteine (NAC). These include:

  * Previous intolerance or allergy to dexamethasone or NAC
  * Scleroderma
  * Active infection
  * Glaucoma
  * Psychiatric disorder that could be exacerbated by dexamethasone
  * Cystinuria
  * Any other condition that the treating physician believes to be a contraindication to dexamethasone or NAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Grade 2-5 Dyspnea within 6 Months Post Radiation Measured by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5 | Up to 6 months post radiation therapy

SECONDARY OUTCOMES:
Patient Scored Dyspnea Measured by Visual Analogue Scale (VAS) | 6 weeks, 3, 6, 9, 12,18, 24, 36, 48, and 60 months post radiation therapy
  Dyspnea (shortness of breath) severity will be reported by participants via a scale, where a score of 100 is no shortness of breath and a score of 0 is the worst shortness of breath ever.
Patient Scored Cough Measured by Visual Analogue Scale (VAS) | 6 weeks, 3, 6, 9, 12,18, 24, 36, 48, and 60 months post radiation therapy
  Cough severity will be reported by participants via a scale, where a score of 100 is no cough and a score of 0 is the worst cough ever.
Quality of Life Measured by FACIT.org Functional Assessment of Cancer Therapy - Lung (FACT-L) Questionnaire | 6 weeks, 3, 6, 9, 12,18, 24, 36, 48, and 60 months post radiation therapy
  The Functional Assessment of Cancer Therapy - Lung (FACT-L ) is a standardized questionnaire used to measure quality of life. The questionnaire consists of 5 scales measuring 37 items in total. Categories of the 5 scales are: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns related to symptoms, cognitive function, and regret of smoking. The score for each item in the scale ranges from 0 to 4, where 0 is not at all and 4 is very much. The scores from each scale are added up, and can be combined to provide a total score.
Quality of Life Measured by EuroQOL Group EQ-5D-5L Questionnaire | 6 weeks, 3, 6, 9, 12,18, 24, 36, 48, and 60 months post radiation therapy
  The EQ-5D-5L is a standardized questionnaire used to measure quality of life and health. The first section includes 5 categories: mobility, self-care, usual activities (e.g. work, family), pain/discomfort, and anxiety/depression. Each category contains 5 statements ranging from no problems to extreme problems, where no problems is assigned a code of 1 and extreme problems is assigned a code of 5. Participants are asked to select the statement that best describes their health that day. No score is generated, rather a 5 digit code is generated based on the response provided, which can then be combined into a data set and interpreted in a variety of ways. The second section includes a 20 cm analogue scale from 0 to 100, where 100 is the best health ever imagined and 0 is the worst health imagined. The participant will mark a score on the scale representing the state of their health on that day.
Local Control as Determined by Radiographic Evidence | 9 years
  Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 will be used to measure tumors in the lung (by size), on imaging, to determine how tumors are responding to treatment.
Progression Free Survival | 9 years
  Time from enrollment to death from any cause or any progression of disease (local, regional, or distant).
Overall Survival | 9 years
  Time from enrollment to death from any cause .
Cancer Specific Survival | 9 years
  Time from enrollment to death from lung cancer, censored at last follow-up or death from other causes.
Rates of Radiation Treatment Completion | 50 months
Rates of Study Drug Completion Rates | 50 months
Rates of Participant Unblinding Related to Adverse Events Development | 50 months

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, Study Chair — London Health Sciences Centre, Lawson Health Research Institute; Houda Bahig, MD, Study Chair — Centre Hospitalier de l'Universite de Montreal
Locations (2):
- Canada (2):
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verstegen NE, Lagerwaard FJ, Hashemi SM, Dahele M, Slotman BJ, Senan S. Patterns of Disease Recurrence after SABR for Early Stage Non-Small-Cell Lung Cancer: Optimizing Follow-Up Schedules for Salvage Therapy. J Thorac Oncol. 2015 Aug;10(8):1195-200. doi: 10.1097/JTO.0000000000000576. PMID 26200274
- [Background] Choi YW, Munden RF, Erasmus JJ, Park KJ, Chung WK, Jeon SC, Park CK. Effects of radiation therapy on the lung: radiologic appearances and differential diagnosis. Radiographics. 2004 Jul-Aug;24(4):985-97; discussion 998. doi: 10.1148/rg.244035160. PMID 15256622
- [Background] Kainthola A, Haritwal T, Tiwari M, Gupta N, Parvez S, Tiwari M, Prakash H, Agrawala PK. Immunological Aspect of Radiation-Induced Pneumonitis, Current Treatment Strategies, and Future Prospects. Front Immunol. 2017 May 2;8:506. doi: 10.3389/fimmu.2017.00506. eCollection 2017. PMID 28512460
- [Background] Tsoutsou PG, Koukourakis MI. Radiation pneumonitis and fibrosis: mechanisms underlying its pathogenesis and implications for future research. Int J Radiat Oncol Biol Phys. 2006 Dec 1;66(5):1281-93. doi: 10.1016/j.ijrobp.2006.08.058. PMID 17126203
- [Background] Niska JR, Schild SE, Rule WG, Daniels TB, Jett JR. Fatal Radiation Pneumonitis in Patients With Subclinical Interstitial Lung Disease. Clin Lung Cancer. 2018 Jul;19(4):e417-e420. doi: 10.1016/j.cllc.2018.02.003. Epub 2018 Feb 17. No abstract available. PMID 29526532
- [Background] Axelsson GT, Putman RK, Aspelund T, Gudmundsson EF, Hida T, Araki T, Nishino M, Hatabu H, Gudnason V, Hunninghake GM, Gudmundsson G. The associations of interstitial lung abnormalities with cancer diagnoses and mortality. Eur Respir J. 2020 Dec 17;56(6):1902154. doi: 10.1183/13993003.02154-2019. Print 2020 Dec. PMID 32646918
- [Background] Ozawa Y, Abe T, Omae M, Matsui T, Kato M, Hasegawa H, Enomoto Y, Ishihara T, Inui N, Yamada K, Yokomura K, Suda T. Impact of Preexisting Interstitial Lung Disease on Acute, Extensive Radiation Pneumonitis: Retrospective Analysis of Patients with Lung Cancer. PLoS One. 2015 Oct 13;10(10):e0140437. doi: 10.1371/journal.pone.0140437. eCollection 2015. PMID 26460792
- [Background] Sanuki N, Ono A, Komatsu E, Kamei N, Akamine S, Yamazaki T, Mizunoe S, Maeda T. Association of computed tomography-detected pulmonary interstitial changes with severe radiation pneumonitis for patients treated with thoracic radiotherapy. J Radiat Res. 2012;53(1):110-6. doi: 10.1269/jrr.110142. PMID 22302051
- [Background] Makimoto T, Tsuchiya S, Hayakawa K, Saitoh R, Mori M. Risk factors for severe radiation pneumonitis in lung cancer. Jpn J Clin Oncol. 1999 Apr;29(4):192-7. doi: 10.1093/jjco/29.4.192. PMID 10340042
- [Background] Lee YH, Kim YS, Lee SN, Lee HC, Oh SJ, Kim SJ, Kim YK, Han DH, Yoo IeR, Kang JH, Hong SH. Interstitial Lung Change in Pre-radiation Therapy Computed Tomography Is a Risk Factor for Severe Radiation Pneumonitis. Cancer Res Treat. 2015 Oct;47(4):676-86. doi: 10.4143/crt.2014.180. Epub 2015 Feb 13. PMID 25687856
- [Background] Yamaguchi S, Ohguri T, Matsuki Y, Yahara K, Oki H, Imada H, Narisada H, Korogi Y. Radiotherapy for thoracic tumors: association between subclinical interstitial lung disease and fatal radiation pneumonitis. Int J Clin Oncol. 2015 Feb;20(1):45-52. doi: 10.1007/s10147-014-0679-1. Epub 2014 Mar 11. PMID 24610080